CLINICAL TRIAL: NCT04401709
Title: A Randomized, Multi-center Phase III Trial of Adjuvant Chemotherapy With Gemcitabine and Capecitabine Compared to Capecitabine Alone in Curatively Resected Biliary Tract Cancer
Brief Title: Gemcitabine+ Capecitabine Vs Capecitabine in Curatively Resected Biliary Tract Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, Principal Investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-01-101
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine/Capecitabine (Experimental): gemcitabine1,000 mg/m2 over 30 min D1, D8, D15 capecitabine 1660 mg/m2, D1-21
  Interventions: Drug: Gemcitabine/Capecitabine
- Capecitabine (Active Comparator): capecitabine 2,500 mg/m2 D1-14
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine/Capecitabine — gemcitabine 1,000 mg / m2 IV on day 1, 8, and 15 of each cycle Capecitabine 1,660mg / m2 PO twice daily 1 ~ 21 days for 4 weeks
  Arms: Gemcitabine/Capecitabine
Drug: Capecitabine — total 8 cycles Capecitabine 1,250 mg / m2 PO twice daily 1 ~ 14 days for 3 weeks
  Arms: Capecitabine

SUMMARY:
This clinical trial is an open-label, multicenter, phase 3 clinical trial to study the efficacy and safety of adjuvant gemcitabine + capecitabine combination treatment in patients with resectable biliary tract cancer according to imaging studies after surgery. All the patients must complete a consent forms before participating in the clinical trial, and the estimated enrollment period is 36 months after IRB approval.

Drug Dose and Schedule:

* Cohort 1: Gemcitabine/Capecitabine, every 4 weeks, total 6 cycles gemcitabine1,000 mg/m2 over 30 min D1, D8, D15 capecitabine 1660 mg/m2, D1-21
* Cohort 2: Capecitabine, everu 3 weeks, total 8 cycles capecitabine 2,500 mg/m2 D1-14

DETAILED DESCRIPTION:
1. Study Background & Rationale:adjuvant capecitabine monotherapy following surgery is regarded as standard treatment after phase 3 BILCAP trial, we need further phase 3 clinical trials to evaluate efficacy of doublet combination adjuvant chemotherapy for Biliary Track Cancer after surgery. Since Korea has much higher incidence rate of Biliary Track Cancer compared to western countries, Korea is considered to be a region that can lead large-scale Biliary Track Cancer clinical trials. In this background, we intend to conduct a randomized phase 3 study to compare adjuvant gemcitabine+cisplatin combination therapy with camecitabine monotherapy following curative intent surgical resection in patients with Biliary Track Cancer .
2. Primary Objective:

   * Disease-free survival at 24 months (2-year DFS)
3. Primary Hypothesis:

   Adjuvant gemcitabine and capecitabine combination treatment confers diseae free survival benefit over capecitabine monotherapy after curative intent surgical resection of biliary tract cancer
4. Study Design:

This clinical trial is an open-label, multicenter, phase 3 clinical trial to study the efficacy and safety of adjuvant gemcitabine + capecitabine combination treatment in patients with resectable biliary tract cancer according to imaging studies after surgery. All the patients must complete a consent forms before participating in the clinical trial, and the estimated enrollment period is 36 months after IRB approval.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed adenocarcinoma of biliary tract canacer (intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder cancer) after curative intent R0 or R1 surgical resection
2. Pathologic disease stage of T2-4, N0-2, M0 after surgery, according to AJCC 8th TNM staging
3. Patients who complete resection (R0 or R1 resection) for biliary tract cancer within 12 weeks of the adjuvant chemotherapy
4. No distant metastasis
5. ECOG performance sstatus score of 0 or 1
6. Age 19 years or older
7. Adequate bone marrow fuction (neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L and hemoglobin ≥9 g/dL)
8. Adequate liver function (total bilirubin < 1.5 fold the upper limit of normal of the study site (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5.0 x ULN)
9. Adequate kidney function (Creatinine < 1.5 x ULN)
10. Unresolved systemic active infection (except for chronic viral hepatitis taking antiviral drugs)
11. Not receiving other drugs for clinical trials or chemotherapy within 30 days prior to randomization
12. A female participant who is not post-menopausal or amenorrhea less than 12 consecutive months without specific reasons is eligible to participate if she is not pregnant, confirmed by serum tests within 7 days before the initiation of chemotherapy
13. The participants provide written informed consent for the study.
14. No prior chemotherapy for biliary tract cancer
15. Participants of childbearing potential must agree to use an adequate method of contraception for the course of the study throught 120 days after the last dose of chemotherapy (oral contraceptives or mechanical contraception such as intrauterine devices or contraceptive barriers and etc). Childbearing potential female is who is not post-menopausal or amenorrhea less than 12 consecutive months without specific reasons

Exclusion Criteria:

1. Other histology type than adenocarcinoma (such as HCC-CCC mixed type or neuroendocrine tumor)
2. Ampula of vater cancer
3. Has known additional malignancy (participants with non-melanoma skin cancer, or carcinoma in situ (e.g. breast carcinoma, prostate cancer) that have undergone potentially curative therapy without recurrence for more than 3 years are not excluded)
4. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
5. Has an active infection requiring systemic therapy (bacteria, virus, fungal, etc)
6. Has a known history of Human Immunodeficiency Virus (HIV)
7. Has an active of hepatitis A or B (patients under anti-B-viral treatment with HBV DNA 1000≤copies/ml is allowed to particiapte).
8. Has a history of severe hemorrhage (gastrointestinal or neurologic) within 2 weeks prior randomization
9. Is unable to take oral drug due to gastrointestinal obstruction or any other conditions.
10. Any history of significant cardiac disease within 3 months prior to randomization including unstable angina, NYHA (The New York Heart Association )III or IV congestive heart failure, myocardiac infarction, or severe uncontrolled arrhythmias
11. Pregnant, breast-feeding or pregnancy test positive female patients
12. Has any contraindications for investigational drug

    * History of hypersensitivity to capecitabine or gemcitabine
    * Any hypersensitivity to fluorouracil drugs
    * Concurrent administration with sorivudine or brivudine
    * DPD(dihydro-pyridine dehydrogenase) deficiency
    * History of TS-1(tegafur / gimeracil / oteracil) administration
    * Galactose intolerance, Lapp lactase deficince, glucose-galactose malabsorption
    * Interstitial pneumonia or pulmonary fibrosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Two-year disease free survival (DFS) | 24 months later

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months later

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea